CLINICAL TRIAL: NCT05063162
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 3, Pivotal Study With an Open-Label Extension Period to Evaluate the Efficacy and Safety of Rozanolixizumab in Adult Participants With Myelin Oligodendrocyte Glycoprotein (MOG) Antibody-Associated Disease (MOG-AD)
Brief Title: A Study to Evaluate the Efficacy and Safety of Rozanolixizumab in Adult Participants With Myelin Oligodendrocyte Glycoprotein (MOG) Antibody-associated Disease (MOG-AD)
Acronym: cosMOG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOG001; 2021-000352-19 (EudraCT Number); 2023-509237-39 (Registry Identifier: EU Clinical Trials); U1111-1301-0122 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease (MOG-AD)
Keywords: MOG; MOGAD; Rozanolixizumab; Myelin oligodendrocyte glycoprotein; Myelin oligodendrocyte glycoprotein antibody-associated disease
MeSH Terms: conditions — Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease | interventions — rozanolixizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: MOG001 consists of a Double-Blind (Part A) and an Open-Label Extension Study Period (Part B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rozanolixizumab Arm (Experimental): Participants randomized into this arm will receive rozanolixizumab at pre-specified timepoints.
  Interventions: Drug: Rozanolixizumab
- Placebo Arm (Placebo Comparator): Participants randomized into this arm will receive placebo at pre-specified timepoints to maintain the blinding.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rozanolixizumab — * Pharmaceutical form: Solution for infusion
  * Route of administration: subcutaneous infusion
  Participants will receive pre-specified doses of rozanolixizumab.
  Other Names: UCB7665
  Arms: Rozanolixizumab Arm
Other: Placebo — * Pharmaceutical form: Solution for infusion
  * Route of administration: subcutaneous infusion
  Participants will receive placebo.
  Other Names: PBO
  Arms: Placebo Arm

SUMMARY:
The purpose of the study is to evalute the efficacy, safety and tolerability of rozanolixizumab for treatment of adult participants with myelin oligodendrocyte glycoprotein (MOG) antibody-associated disease (MOG-AD).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 to ≤89 years of age, at the time of signing the informed consent
* Confirmed diagnosis of MOG-AD consistent with published diagnostic criteria for MOG-AD
* Participant has history of relapsing MOG-AD with at least 1 documented relapse over the last 12 months and a documented positive serum MOG Ab test using a cell-based assay (CBA) within 6 months prior to randomization
* Participant must be clinically stable at the time of the Screening Visit and during the Screening Period

Exclusion Criteria:

* Participant has been diagnosed with a neurological autoimmune disease (including multiple sclerosis (MS) and aquaporin-4 positive neuromyelitis optica spectrum disorder (NMOSD)), or a systemic autoimmune disease that in the opinion of the investigator can interfere with the safety of the participant
* Participant has a clinically important active infection (including unresolved or not adequately treated infection) as assessed by the investigator, including participants with a serious infection within 6 weeks prior to the first dose of the investigational medicinal product (IMP)
* Participant has a current or medical history of primary immunodeficiency
* Participant tests positive for aquaporin-4 antibodies at Screening
* Participant has a serum total IgG level ≤ 5.5g/L

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2027-05-06 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
For Part A: Time from randomization to first independently centrally adjudicated relapse (TTFR) during the DB Treatment Period | Baseline (Week 1) to EDB/EWD Visit (until a confirmed relapse or up to approximately 132 weeks)
  The TTFR (days) will be defined as the interval between the date of randomization and the first date of the objective relapse.
  During the Double Blind (DB) Treatment Period (Part A); EDB/EWD = End of Double-Blind/Early Withdrawal Visit
For Part B: Incidence of treatment-emergent adverse events (TEAEs) during OLE Treatment Period | OLE Treatment Period (OLE Week 1) to EOS/EWD Visit (up to OLE Week 52)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP.
  Open-Label Extension (OLE) Treatment Period (Part B); EOS/EWD = End of Study/Early Withdrawal Visit.
For Part B: Incidence of treatment-emergent adverse events (TEAEs) leading to permanent withdrawal of investigational medicinal product (IMP) during OLE Treatment Period | OLE Treatment Period (OLE Week 1) to EOS/EWD Visit (up to OLE Week 52)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs leading to discontinuation of the study are reported.
  During Part B.

SECONDARY OUTCOMES:
For Part A: Change from Baseline in Low-Contrast Monocular Visual Acuity (Worst Affected Eye) measured by low-contrast Landolt C Broken Rings Chart at the EDB/EWD Visit | From Baseline (Week 1) to EDB/EWD Visit (until a confirmed relapse or up to approximately 132 weeks)
  Visual acuity is a measurement of the capacity for visual discrimination of fine details. Visual acuity tests are used to determine the smallest characters that can be read on a standardized chart. The Landolt C Broken Ring Chart uses standardized incomplete rings or "C", which are positioned in any direction in the chart (up, down, left, right, and 45 degree positions in between). The participant has to be able to indicate where the break of the "C" is located, by describing the position or by giving gesture.
  During Part A.
For Part A: Disability as assessed by Expanded Disability Status Scale (EDSS) scores at the EDB/EWD Visit (with confirmation at 3 months) | Baseline (Week 1), EDB/EWD Visit (until a confirmed relapse or up to approximately 132 weeks)
  The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death) in half-point increments with half steps from 1.0 to 9.5. The higher the value the higher is the level of impairment and disability.
  During Part A.
For Part A: Number of MOG-AD related inpatient hospitalizations during the DB Treatment Period | Baseline (Week 1) to EDB/EWD Visit (until a confirmed relapse or up to approximately 132 weeks)
  The total number of MOG-AD related hospitalizations from Baseline through EDB/EWD Visit.
  During Part A.
For Part A: Incidence of treatment-emergent adverse events (TEAEs) during the DB Treatment Period | Baseline (Week 1) to EDB/EWD Visit (until a confirmed relapse or up to approximately 132 weeks)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP.
  During Part A.
For Part B: Independently centrally adjudicated annualized relapse rate (ARR) during the DB and OLE Treatment Period | Baseline (Week 1) to EOS/EWD Visit (up to OLE Week 52)
  An ARR will be calculated for each participant prior to randomization into the Double-Blind Treatment Period (based on available historical data), and 2 ARRs after randomization to study treatment: first for relapses occurring during the Double-Blind Treatment Period and the second for relapses occurring during the OLE Treatment Period. The relapse episodes for each participant will be recorded throughout the entire study.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (83):
- United States (15):
  - Mog001 50297, Scottsdale, Arizona
  - Mog001 50450, Palo Alto, California
  - Mog001 50101, Aurora, Colorado
  - Mog001 50553, Washington D.C., District of Columbia
  - Mog001 50342, Jacksonville, Florida
  - Mog001 50308, Tampa, Florida
  - Mog001 50472, Peoria, Illinois
  - Mog001 50074, Kansas City, Kansas
  - Mog001 50552, Baltimore, Maryland
  - Mog001 50243, Boston, Massachusetts
  - Mog001 50104, Rochester, Minnesota
  - Mog001 50571, Cleveland, Ohio
  - Mog001 50304, Dallas, Texas
  - Mog001 50568, San Antonio, Texas
  - Mog001 50473, Salt Lake City, Utah
- Australia (2):
  - Mog001 30022, Melbourne
  - Mog001 30026, Southport
- Belgium (4):
  - Mog001 40123, Anderlecht
  - Mog001 40756, Bruxelles/brussel
  - Mog001 40122, Edegem
  - Mog001 40185, Ghent
- Mog001 60033, Porto Alegre, Brazil
- Czechia (3):
  - Mog001 40195, Hradec Králové
  - Mog001 40124, Prague
  - Mog001 40721, Teplice
- France (5):
  - Mog001 40657, Bron
  - Mog001 40422, Caen
  - Mog001 40130, Marseille
  - Mog001 40755, Montpellier
  - Mog001 40170, Strasbourg
- Germany (5):
  - Mog001 40659, Berlin
  - Mog001 40386, Cologne
  - Mog001 40140, Göttingen
  - Mog001 40177, Münster
  - Mog001 40577, Ulm
- Greece (2):
  - Mog001 40850, Athens
  - Mog001 40851, Thessaloniki
- Italy (3):
  - Mog001 40146, Pavia
  - Mog001 40629, Roma
  - Mog001 40646, Verona
- Japan (10):
  - Mog001 20225, Bunkyō City
  - Mog001 20068, Chiba
  - Mog001 20307, Isehara
  - Mog001 20049, Kitakyushu
  - Mog001 20143, Kodaira
  - Mog001 20223, Kōriyama
  - Mog001 20224, Sendai
  - Mog001 20227, Sendai
  - Mog001 20070, Shinjuku-ku
  - Mog001 20032, Suita
- Mexico (2):
  - Mog001 50486, Culiacán
  - Mog001 50485, Mexico City
- Mog001 40840, Bydgoszcz, Poland
- Portugal (2):
  - Mog001 40485, Coimbra
  - Mog001 40669, Porto
- South Korea (2):
  - Mog001 20226, Goyang-si
  - Mog001 20104, Seoul
- Spain (6):
  - Mog001 40267, Barcelona
  - Mog001 40100, Madrid
  - Mog001 40161, Madrid
  - Mog001 40341, Málaga
  - Mog001 40350, Murcia
  - Mog001 40049, Seville
- Sweden (2):
  - Mog001 40660, Gothenburg
  - Mog001 40663, Huddinge
- Switzerland (3):
  - Mog001 40723, Basel
  - Mog001 40337, Bern
  - Mog001 40630, Zurich
- Taiwan (6):
  - Mog001 20096, Changhua
  - Mog001 20303, Kaohsuing CITY
  - Mog001 20080, Taichung
  - Mog001 20094, Tainan
  - Mog001 20304, Taipei
  - Mog001 20082, Taoyuan
- Turkey (Türkiye) (5):
  - Mog001 40849, Bursa
  - Mog001 40550, Istanbul
  - Mog001 40726, Izmir
  - Mog001 40648, Samsun
  - Mog001 40725, Sancaktepe
- Ukraine (2):
  - Mog001 20319, Kyiv
  - Mog001 20228, Ternopil
- United Kingdom (2):
  - Mog001 40661, Liverpool
  - Mog001 40163, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Derived] Mader S, Kumpfel T, Meinl E. Pathomechanisms in demyelination and astrocytopathy: autoantibodies to AQP4, MOG, GFAP, GRP78 and beyond. Curr Opin Neurol. 2022 Jun 1;35(3):427-435. doi: 10.1097/WCO.0000000000001052. PMID 35674086